CLINICAL TRIAL: NCT03330795
Title: Bilateral Orthotopic Lung Transplant in Tandem With CD3+ and CD19+ Cell Depleted Bone Marrow Transplant From Partially HLA Matched Cadaveric Donors (RTB-003)
Brief Title: Bilateral Orthotopic Lung Transplant - Bone Marrow Transplant
Acronym: BOLT-BMT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Pittsburgh (Other); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT BOLT-BMT; DAIT RTB-003 (Other: NIAID, NIH); U01AI125050 (NIH); NIAID DAIT CRMS ID#: 32935 (Other: DAIT NIAID)
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Primary Immunodeficiency; PID
Keywords: end-stage lung disease; Bilateral Orthotopic Lung Transplant (BOLT) candidate; CD3/CD19 negative allogeneic hematopoietic stem cells (HSCT); CD3+/CD19+ depleted Bone Marrow Transplant (BMT); Cadaveric (Deceased) Donor; Unrelated (Deceased) Donor
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CD3/CD19 neg allogeneic BMT (Experimental): Participants may receive a double lung transplant followed by a bone marrow (hematopoietic stem cells) transplant, if a partially HLA-matched organ offer is accepted. The lungs and allogeneic hematopoietic stem cells will be from the same partially HLA-matched cadaveric donor. Prior to marrow transplantation, the marrow will be negatively selected for CD3/CD19 using a CliniMACS® depletion device.
  Interventions: Biological: CD3/CD19 neg allogeneic BMT

INTERVENTIONS:
Biological: CD3/CD19 neg allogeneic BMT — Negative selection for CD3/CD19 will be performed on a CliniMACS® depletion device within 36 hours of collection, and cryopreserved for later marrow transplantation. BMT conditioning and transplantation will start at least 8 weeks or more post lung transplant - once the participant is clinically judged suitable to undergo BMT conditioning and transplantion.
  Other Names: CD3+/CD19+ depleted HSCT

SUMMARY:
The purpose of this study is to determine whether bilateral orthotopic lung transplantation (BOLT) followed by cadaveric partially-matched CD3+/CD19+ depleted bone marrow transplant (BMT) is safe and effective for individuals aged 10 through 45 years with the diagnosis of primary immunodeficiency (PID) and end-stage lung disease.

The enrollment goal: 8 participants who receive both BOLT and BMT.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the safety and efficacy of performing bilateral orthotopic lung transplantation (BOLT) followed by cadaveric, partially HLA-matched CD3+/CD19+-depleted hematopoietic stem cell transplantation (HSCT) from the same donor for participants with primary immunodeficiency diseases (PID) and end-stage lung disease. For many patients with primary immunodeficiencies, HSCT, which we refer to as Bone Marrow Transplant (BMT) is a curative, life-saving therapy, resulting in restoration of function in the immune system. Patients with primary immunodeficiencies often develop pulmonary complications as a result of chronic or recurrent infections, making them ineligible for BMT due to the high risk of mortality and pulmonary complications. Lung transplant prior to BMT would allow for restoration of pulmonary function prior to BMT, allowing PID patients to proceed to BMT , which would be curative for the patient's underlying immunodeficiency. As a secondary aim, after successful engraftment with donor bone marrow, the feasibility of participants tolerating planned withdrawal of immunosuppression and achieving eventual freedom from all immunosuppressive drugs and attaining a tolerant state will be assessed.

This is a single center study in which participants receive a cadaveric, partially Human Leukocyte Antigen (HLA)-matched lung transplant followed by a CD3+/CD19+ depleted bone marrow transplant (BMT) from the same donor. In this study, the investigators will use a ≥ 2/6 HLA-matched T cell depleted bone marrow transplant from a cadaveric organ donor with an identical ABO blood type as the recipient.

Participants will undergo:

* Bilateral orthotopic lung transplant (BOLT) utilizing basiliximab induction or an alternate induction therapy based on their underlying disease. Rituximab may be initiated prior to the lung transplant, with tacrolimus as the ongoing maintenance immunosuppression.
* BMT utilizing CD3+/CD19+-depleted bone marrow with bone marrow conditioning beginning no less than 8 weeks after BOLT.

The duration of participant involvement in the trial is up to 2 years post-BMT.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or parent guardian must be able to understand and provide informed consent;
* Subject fulfills criteria for United Network of Organ Sharing (UNOS) listing;
* Subject must have evidence of an underlying primary immunodeficiency for which Bone Marrow Transplant (BMT) is clinically indicated. Examples of such diseases include, but are not limited to:

  * Severe Combined Immunodeficiency (SCID)
  * Combined immunodeficiency with defects in T-cell-mediated immunity, including Omenn syndrome and DiGeorge Syndrome
  * Severe Chronic Neutropenia
  * Chronic Granulomatous Disease (CGD)
  * Hyper Immunoglobulin E (IgE) Syndrome or Job's Syndrome
  * CD40 or CD40L deficiency
  * Wiskott-Aldrich Syndrome
  * Mendelian Susceptibility to Mycobacterial Disease
  * GATA2-associated Immunodeficiency.
* Subjects must have evidence of end-stage lung disease and be candidates for bilateral orthotopic lung transplant as determined by the lung transplant team;
* Glomerular filtration rate (GFR) ≥ 50 mL/min/1.73 m^2;
* Aspartate aminotransferase (AST), Alanine aminotransaminase (ALT) ≤ 4x upper limit of normal, total bilirubin ≤ 2.5 mg/dL, normal INR;
* Cardiac ejection fraction ≥ 40% or shortening fraction ≥ 26%;
* Negative pregnancy test for females >10 years old or who have reached menarche, unless surgically sterilized;
* All females of childbearing potential and sexually active males must agree to use a Food and Drug Administration (FDA) approved method of birth control for up to 24 months after BMT or for as long as they are taking any medication that may harm a pregnancy, an unborn child or may cause birth defect; and
* Subject and/or parent guardian will also be counseled regarding the potential risks of infertility following BMT and advised to discuss sperm banking or oocyte

  * harvesting.

Eligibility for Bone Marrow Transplant*:

* GFR >50 mL/min/1.73 m^2;
* AST, ALT <4x upper limit of normal, Total bilirubin < 2.5 mg/dL;
* Cardiac ejection fraction ≥40% or shortening fraction of at least 26%;
* Human Immunodeficiency Virus (HIV) negative by serology and PCR;
* Human T-lymphotropic virus (HTLV) serology negative;
* Forced vital capacity (FVC) and Forced expiratory volume (FEV1) ≥ 40% predicted for age and SpO2 of >90% at rest on room air AND with clearance by the lung transplant team;
* Absence of uncontrolled infection as determined by blood cultures and radiographic results of previously affected sites, in particular, pulmonary densities during the past 2 weeks prior to chemotherapy;
* Absence of Acute Cellular Rejection (ACR); and
* Bone marrow processing has been completed, and an appropriate stem cell product is available for administration.

  * Note: The decision to proceed with the BMT will be at the discretion of the lung transplant team following clearance by the bone marrow team based on the criteria below. The conditioning for the BMT will begin no less than 8 weeks following the lung transplant.

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol;
* Subjects who have underlying malignant conditions;
* Subjects who have non-malignant conditions that do not require hematopoietic stem cell transplantation;
* Human Immunodeficiency Virus (HIV) positive by serology or polymerase chain reaction (PCR), human T-lymphotropic virus (HTLV) positive by serology;
* Females who are pregnant or who are lactating;
* Allergy to dimethyl sulfoxide (DMSO) or any other ingredient used in the manufacturing of the stem cell product;
* Uncontrolled pulmonary infection, as determined by radiographic findings and/or significant clinical deterioration.

  -- Pulmonary colonization with multiple organisms is common, and will not be considered an exclusion criterion.
* Uncontrolled systemic infection, as determined by the appropriate confirmatory testing e.g. blood cultures, PCR testing, etc.;
* Recent recipient of any licensed or investigational live attenuated vaccine(s), within 4 weeks of transplant; or
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose:

  * additional risks from participation in the study,
  * may interfere with the participant's ability to comply with study requirements,
  * or that may impact the quality or interpretation of the data obtained from the study.

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Szabolcs, MD, Study Chair — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- BOLT-BMT Protocol: Participants may receive a double lung transplant followed by a bone marrow (hematopoietic stem cells) transplant, if a partially HLA-matched organ offer is accepted. The lungs and allogeneic hematopoietic stem cells will be from the same partially HLA-matched cadaveric donor. Prior to marrow transplantation, the marrow will be negatively selected for CD3/CD19 using a CliniMACS® depletion device.
  CD3/CD19 neg allogeneic BMT: Negative selection for CD3/CD19 will be performed on a CliniMACS® depletion device within 36 hours of collection, and cryopreserved for later marrow transplantation. BMT conditioning and transplantation will start at least 8 weeks or more post lung transplant - once the participant is clinically judged suitable to undergo BMT conditioning and transplantion.
Period: Overall Study
Arm/Group | BOLT-BMT Protocol
Started | 5
Completed | 1
Not Completed | 4
Not completed — Death | 3
Not completed — No longer eligible to receive transplants or study interventions due to medical contraindication | 1

BASELINE CHARACTERISTICS:
Arm/Group | BOLT-BMT Protocol
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Primary Immunodeficiency [Number; unit: Participants]
  B-cell disorder (e.g. CVID) | 2
  T-cell lymphopenia/T-cell disorder (SCID, CID) | 2
  Myeloid disorder (e.g. CGD) | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety: Death
Description: How many, if any, participants die during study participation.
Time Frame: Average of approximately 31 months for those who received an initial transplant
Population: This Number of Participants analyzed includes one participant who became ineligible: no longer eligible to receive transplants or study interventions due to medical contraindication. One participant was terminated from the study prior to receiving a study transplant, prior to developing fatal illness, because this patient developed an infection which made her ineligible to proceed to transplant. This participant died during follow-up of safety events on study after termination from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | BOLT-BMT Protocol
Number analyzed (Participants) | 5
Participants | 4

2. Primary Outcome: Safety: Engraftment Syndrome
Description: How many, if any, participants develop engraftment syndrome.
Time Frame: Average of ~7.5 months of time post BMT for those receiving both lung and BMT transplants.
Population: Recipients of CD3/CD19-depleted marrow
Measure: Count of Participants; unit: Participants
Groups:
- CD3/CD19 Neg Allogeneic BMT: Participants who received a bilateral lung transplant and subsequently received a CD3/CD19 depleted marrow transplant.
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 3
Participants | 0

3. Primary Outcome: Engraftment Failure
Time Frame: Average of ~7.5 months of time post BMT for those receiving both lung and BMT transplants.
Population: Recipients of CD3/CD19-depleted marrow
Measure: Count of Participants; unit: Participants
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 3
Participants | 1

4. Primary Outcome: Grade 4 or 5 Events Potentially Attributable to Rituximab
Time Frame: Average of ~25 months.
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | BOLT-BMT Protocol
Number analyzed (Participants) | 5
Participants | 4

5. Primary Outcome: BOS at 1 Year Post BOLT
Description: Diagnosis of BOS (Bronchiolitis Obliterans Syndrome) at any time up to 1 year post BOLT. BOS is one of the undesirable complications of lung transplantation.
Time Frame: throughout the first year post BOLT
Population: Recipients of CD3/CD19-depleted marrow (includes 1 participant receiving BMT >1 year post BOLT)
Measure: Count of Participants; unit: Participants
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 3
Participants | 0

6. Primary Outcome: Efficacy: Count of Participants With Requirement for Supplemental Oxygen and/or Ventilatory Support
Description: The number of participant(s) who need either supplemental oxygen and/or ventilator support (noninvasive/invasive) will be assessed using the Bronchiolitis Obliterans Syndrome (BOS) Classification Score for pulmonary function (e.g., the Forced Expiratory Volume in 1 Second (FEV1). FEV1 is air volume exhaled in 1 second during spirometry, a lung function test. (Continuing dependence on supplemental oxygen or ventilatory support is an undesirable outcome of lung transplantation).
Time Frame: at 1 Year Post Lung Transplant (BOLT)
Population: Recipients of CD3/CD19-depleted marrow (includes 1 participant receiving BMT >1 year post BOLT)
Measure: Count of Participants; unit: Participants
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 3
Participants | 0

7. Primary Outcome: Efficacy: Count of Participants With T-cell Chimerism
Description: The number of participants who have ≥ 25% donor T-cell chimerism.
Time Frame: 1 Year Post Bone Marrow Transplant (BMT)
Population: Recipients of CD3/CD19-depleted marrow
Measure: Count of Participants; unit: Participants
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 3
Participants | 1

8. Primary Outcome: Efficacy: Count of Participants With Myeloid Chimerism
Description: The number of participants with myeloid disorders (e.g. Chronic Granulomatous Disease [CGD]) who attain ≥ 10% myeloid chimerism.
Time Frame: 1 Year Post Bone Marrow Transplant (BMT)
Population: Recipients of CD3/CD19-depleted marrow
Measure: Count of Participants; unit: Participants
Groups:
- CD3/CD19 Neg Allogeneic BMT: Participants with PID myeloid disorder who received a bilateral lung transplant and subsequently received a CD3/CD19 depleted marrow transplant.
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 1
Participants | 1

9. Primary Outcome: Efficacy: Count of Participants B-cell Chimerism
Description: The number of participants with B-cell disorders who attain ≥ 10% B-cell chimerism.
Time Frame: 1 Year Post Bone Marrow Transplant (BMT)
Population: Recipients of CD3/CD19-depleted marrow
Measure: Count of Participants; unit: Participants
Groups:
- CD3/CD19 Neg Allogeneic BMT: Participants with a PID B-cell disorder who received a bilateral lung transplant and subsequently received a CD3/CD19 depleted marrow transplant.
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 2
Participants | 0

10. Secondary Outcome: Count of Participants Able to Proceed to BMT
Description: The number of participants for which it is feasible to proceed to BMT within 6 months following lung transplant.
Time Frame: 6 Months Post Lung Transplant (BOLT)
Population: Recipients of a bilateral lung transplant
Measure: Count of Participants; unit: Participants
Groups:
- Lung Transplant: Participants who received a bilateral lung transplant.
Arm/Group | Lung Transplant
Number analyzed (Participants) | 4
Participants | 1

11. Secondary Outcome: Count of Participants Who Achieve Tolerance
Description: The number of participants who develop tolerance to both the host and pulmonary graft.
  Definition of tolerance: A participant's successful withdrawal from systemic immunosuppression for 6 weeks with no increase cGVHD score and stable or improving PFTs.
Time Frame: Average of ~7.5 months of time post BMT for those receiving both lung and BMT transplants.
Population: Recipients of CD3/CD19-depleted marrow
Measure: Count of Participants; unit: Participants
Groups:
- CD3/CD19 Neg Allogeneic BMT: Participants who received bilateral lung transplant and subsequently received the CD3/CD19 depleted marrow transplant.
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 3
Participants | 0

12. Secondary Outcome: Long Term Complications of Combined Solid Organ and Bone Marrow Transplant
Description: Summary of long-term complications of combined solid organ and bone marrow transplant (BMT).
Time Frame: Average of ~7.5 months of time post BMT for those receiving both lung and BMT transplants.
Population: Recipients of CD3/CD19-depleted marrow
Measure: Count of Participants; unit: Participants
Groups:
- CD3/CD19 Neg Allogeneic BMT: Participants who received a bilateral lung transplant and subsequently received the CD3/CD19-depleted marrow transplant.
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 3
Participants | 0

13. Secondary Outcome: Count of Participants Who Develop Acute Cellular Rejection and Graft Failure
Description: The number of participants who develop acute cellular rejection and graft failure post BMT.
Time Frame: Average of ~7.5 months of time post BMT for those receiving both lung and BMT transplants.
Population: Recipients of CD3/CD19-depleted marrow
Measure: Count of Participants; unit: Participants
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 3
Participants | 0

14. Secondary Outcome: Count of Participants Able to Initiate Withdrawal of Immunosuppression
Description: The number of participants who are able to start immunosuppression withdrawal.
Time Frame: 1 year following BMT
Population: Recipients of CD3/CD19-depleted marrow
Measure: Count of Participants; unit: Participants
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 3
Participants | 0

15. Secondary Outcome: Time to Withdrawal of Immunosuppression
Description: Time from BMT to withdrawal of immunosuppression.
Time Frame: Average of ~7.5 months of time post BMT for those receiving both lung and BMT transplants.
Population: None of the participants withdrew from IS during study participation.
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 0

16. Secondary Outcome: Time to Independence From Treatment Dose Antimicrobial Drug
Description: A measure of pathogen-specific immunity.
Time Frame: Average of ~7.5 months of time post BMT for those receiving both lung and BMT transplants.
Population: None of the participants achieved independence from treatment dose antimicrobial drugs during study participation.
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 0

17. Secondary Outcome: Post-BMT Achievement of Normal Lymphocyte Count for T-cell Lymphopenias
Description: For participants with immune deficiencies with T cell lymphopenias, number of participants achieving age adjusted, low limit normal range lymphocyte count by 1-year post-BMT.
Time Frame: 1 year post BMT
Population: Recipients of CD3/CD19-depleted marrow
Measure: Count of Participants; unit: Participants
Groups:
- CD3/CD19 Neg Allogeneic BMT: Participants with a PID of T-cell disorder/T-cell lymphopenia who received a bilateral lung transplant and subsequently received the CD3/CD19-depleted marrow transplant.
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 2
Participants | 0

18. Secondary Outcome: Count of Participants Who Develop Acute Graft-Versus-Host Disease (GVHD)
Description: The number of participants who develop acute graft-versus-host disease (GVHD) following tandem BOLT and BMT.
Time Frame: Average of ~7.5 months of time post BMT for those receiving both lung and BMT transplants.
Population: Recipients of CD3/CD19-depleted marrow
Measure: Count of Participants; unit: Participants
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 3
Participants | 1

19. Secondary Outcome: Count of Participants With Chronic Graft-Versus-Host Disease (GVHD)
Description: The number of participants who develop chronic graft-versus-host disease (GVHD) following tandem BOLT and BMT.
Time Frame: Average of ~7.5 months of time post BMT for those receiving both lung and BMT transplants.
Population: Recipients of CD3/CD19-depleted marrow
Measure: Count of Participants; unit: Participants
Arm/Group | CD3/CD19 Neg Allogeneic BMT
Number analyzed (Participants) | 3
Participants | 0

20. Secondary Outcome: Count of Participants Who Develop Chronic Lung Allograft Dysfunction or Allograft Failure
Description: A significant development in chronic lung allograft dysfunction (as evidenced by a change in BOS stage) or allograft failure at 1 year and up to 2 year post lung transplant (for lung transplant alone and BOLT-BMT subjects.
Time Frame: up to 2 years post BOLT
Population: Recipients of a bilateral lung transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Lung Transplant
Number analyzed (Participants) | 4
Participants | 0

21. Secondary Outcome: Count of Pre-BMT Conditioning Rituximab Related Adverse Events
Description: The number of Grade 4 or 5 adverse events possibly related to the use of rituximab prior to the start of BMT conditioning.
Time Frame: Average of approximately 9 months.
Population: All participants, prior to the start of BMT Conditioning
Measure: Count of Participants; unit: Participants
Groups:
- Pre-conditioning: BOLT-BMT Protocol: Participants may receive a double lung transplant followed by a bone marrow (hematopoietic stem cells) transplant, if a partially HLA-matched organ offer is accepted. The lungs and allogeneic hematopoietic stem cells will be from the same partially HLA-matched cadaveric donor. Prior to marrow transplantation, the marrow will be negatively selected for CD3/CD19 using a CliniMACS® depletion device.
  CD3/CD19 neg allogeneic BMT: Negative selection for CD3/CD19 will be performed on a CliniMACS® depletion device within 36 hours of collection, and cryopreserved for later marrow transplantation. BMT conditioning and transplantation will start at least 8 weeks or more post lung transplant - once the participant is clinically judged suitable to undergo BMT conditioning and transplantion.
Arm/Group | Pre-conditioning: BOLT-BMT Protocol
Number analyzed (Participants) | 5
Participants | 3

ADVERSE EVENTS:
Time Frame: Average of approximately 25 months
Arm/Group | BOLT-BMT Protocol
All-Cause Mortality (participants affected / at risk) | 4/5
Serious Adverse Events (participants affected / at risk) | 5/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOLT-BMT Protocol (N=5)
Acute graft versus host disease in intestine (Immune system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (7)
Bone marrow disorder (Blood and lymphatic system disorders) | 1 (1)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Feeling abnormal (General disorders) | 1 (1)
Fluid balance positive (Investigations) | 1 (1)
Fungal sepsis (Infections and infestations) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2)
Infection (Infections and infestations) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1)
Meningitis (Nervous system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Otitis externa (Ear and labyrinth disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Metabolism and nutrition disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Vascular disorders) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOLT-BMT Protocol (N=5)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (6)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (2)
Acid base balance abnormal (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2)
Acute graft versus host disease in skin (Immune system disorders) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (7)
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Administration related reaction (General disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (6)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Appetite disorder (Metabolism and nutrition disorders) | 1 (1)
Ascites (Hepatobiliary disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Aspergillus infection (Infections and infestations) | 1 (1)
Aspergillus test positive (Investigations) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Bacteraemia (Infections and infestations) | 1 (1)
BK virus infection (Infections and infestations) | 1 (1)
Blood albumin decreased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (3)
Blood bilirubin increased (Investigations) | 2 (4)
Blood calcium decreased (Investigations) | 1 (1)
Blood count abnormal (Investigations) | 1 (2)
Blood creatinine increased (Investigations) | 2 (2)
Blood disorder (Blood and lymphatic system disorders) | 1 (1)
Blood electrolytes decreased (Investigations) | 1 (1)
Blood electrolytes increased (Investigations) | 1 (1)
Blood fibrinogen decreased (Investigations) | 1 (2)
Blood immunoglobulin A decreased (Investigations) | 1 (1)
Blood immunoglobulin G decreased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood magnesium decreased (Investigations) | 2 (2)
Blood magnesium increased (Investigations) | 2 (2)
Blood parathyroid hormone increased (Investigations) | 1 (1)
Blood phosphorus decreased (Investigations) | 2 (2)
Blood potassium decreased (Investigations) | 1 (3)
Blood potassium increased (Investigations) | 3 (5)
Blood pressure decreased (Investigations) | 1 (1)
Blood test abnormal (Investigations) | 2 (2)
Blood triglycerides increased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (1)
Bloody discharge (General disorders) | 1 (1)
Body tinea (Skin and subcutaneous tissue disorders) | 1 (1)
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 1 (1)
Breath sounds abnormal (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (3)
Candida infection (Infections and infestations) | 1 (1)
Cardiogenic shock (Vascular disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Cardiovascular symptom (Cardiac disorders) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (2)
Cerebrovascular disorder (Vascular disorders) | 1 (1)
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest X-ray abnormal (Investigations) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (3)
Clostridium difficile colitis (Gastrointestinal disorders) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 2 (2)
Cognitive disorder (Psychiatric disorders) | 1 (1)
Complication associated with device (General disorders) | 1 (1)
Compression fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Cutaneous symptom (Skin and subcutaneous tissue disorders) | 2 (5)
Dental caries (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diaphragm muscle weakness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (13)
Dizziness (Nervous system disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Endocarditis (Cardiac disorders) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (2)
Enterovirus infection (Infections and infestations) | 1 (1)
Enzyme level increased (Investigations) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Epistaxis (Vascular disorders) | 1 (1)
Epstein-Barr viraemia (Infections and infestations) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Eustachian tube disorder (Ear and labyrinth disorders) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1)
Fibrin D dimer increased (Investigations) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fluid balance negative (Investigations) | 1 (1)
Fluid balance positive (Investigations) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Flushing (General disorders) | 1 (1)
Fungal infection (Infections and infestations) | 3 (4)
Gamma-glutamyltransferase decreased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastroenteritis norovirus (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (General disorders) | 2 (5)
Gastrointestinal inflammation (General disorders) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
General symptom (General disorders) | 2 (4)
Glucose urine present (Investigations) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3)
Haemoglobin decreased (Investigations) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (2)
Hallucination (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (4)
Hepatic enzyme increased (Investigations) | 1 (1)
Hyperammonaemia (Hepatobiliary disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycaemia (Endocrine disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (5)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hyperprothrombinaemia (Blood and lymphatic system disorders) | 1 (2)
Hypertension (Vascular disorders) | 4 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (6)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (5)
Hypothyroidism (Endocrine disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Incontinence (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Investigation abnormal (Investigations) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Laboratory test abnormal (Investigations) | 2 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 4 (5)
Liver function test abnormal (Investigations) | 2 (2)
Liver function test decreased (Investigations) | 1 (1)
Liver function test increased (Investigations) | 2 (2)
Localised oedema (General disorders) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (7)
Lymphoedema (Vascular disorders) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 1 (1)
Medical device site pain (Injury, poisoning and procedural complications) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1)
Monocyte count decreased (Investigations) | 2 (3)
Monocyte count increased (Investigations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Muscle injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Musculoskeletal chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Mycobacterial infection (Infections and infestations) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (10)
Neutrophil count decreased (Investigations) | 3 (5)
Neutrophil count increased (Investigations) | 4 (4)
Nodular regenerative hyperplasia (Hepatobiliary disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (4)
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nonspecific reaction (General disorders) | 1 (1)
Occult blood positive (Investigations) | 1 (1)
Oedema (General disorders) | 2 (2)
Oedema genital (Reproductive system and breast disorders) | 1 (1)
Oedema peripheral (General disorders) | 4 (4)
Oedema peripheral (Metabolism and nutrition disorders) | 2 (3)
Oliguria (Renal and urinary disorders) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (3)
Oral disorder (Gastrointestinal disorders) | 1 (2)
Otitis externa (Ear and labyrinth disorders) | 1 (1)
Pain (General disorders) | 2 (3)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Petechiae (Blood and lymphatic system disorders) | 1 (1)
Pharyngitis streptococcal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Platelet count decreased (Investigations) | 3 (7)
Platelet count increased (Investigations) | 1 (1)
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Postoperative delirium (Psychiatric disorders) | 1 (2)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Protein-losing gastroenteropathy (Gastrointestinal disorders) | 1 (1)
Protein total decreased (Investigations) | 1 (1)
Protein urine (Investigations) | 1 (1)
Protein urine present (Investigations) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary function test decreased (Investigations) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Renal cyst (Renal and urinary disorders) | 1 (1)
Respiratory acidosis (Metabolism and nutrition disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Reticulocyte count decreased (Investigations) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right ventricular systolic pressure increased (Investigations) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin bacterial infection (Skin and subcutaneous tissue disorders) | 1 (2)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (3)
Skin discomfort (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Spinal compression fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Sputum culture positive (Investigations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Temperature regulation disorder (General disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3)
Tremor (Nervous system disorders) | 3 (3)
Ultrasound liver abnormal (Investigations) | 1 (1)
Ultrasound scan abnormal (Investigations) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary casts present (Investigations) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Viral infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (6)
Weight decreased (Investigations) | 1 (1)
Weight loss diet (Surgical and medical procedures) | 1 (1)
White blood cell count decreased (Investigations) | 4 (8)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT03330795/Prot_SAP_000.pdf
  • Informed Consent Form: Adult Informed Consent (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT03330795/ICF_005.pdf
  • Informed Consent Form: Child Informed Consent (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT03330795/ICF_006.pdf